CLINICAL TRIAL: NCT00656162
Title: Ultrasound Detection of Radiographically Negative Fractures of Elbow in Children
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: SIM005-HMO-CTILL
Record Dates: First submitted 2008-04-06; First posted 2008-04-10 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-10

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Fractures of an elbow are common in children. Accurate initial diagnosis is crucial for the management of the fractures of an elbow. In young children the fractures may be suspected clinically but missed on x-rays due to mostly non-ossified cartilage that is not visible on a regular x-ray. We propose that every x-ray negative, but clinically suspicious elbow trauma in children can be additionally evaluated using high resolution US.

ELIGIBILITY:
Inclusion Criteria:

* Signing Informed consent

Exclusion Criteria:

* Unwillingness to sign informed consent.
* Any fracture of the same hand or forearm before or after an avaluated event.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with clinically suspected but x-ray negative elbow trauma
Sampling Method: Non-Probability Sample
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel